CLINICAL TRIAL: NCT02267525
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Phase 2 Study to Assess the Efficacy, Safety, and Tolerability of Velusetrag for the Treatment of Diabetic or Idiopathic Gastroparesis
Brief Title: The Diabetic and Idiopathic Gastroparesis Efficacy, Safety, and Tolerability (DIGEST) Study
Acronym: DIGEST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Collaborators: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0099
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Gastroparesis
Keywords: Gastroparesis; Diabetic; Idiopathic
MeSH Terms: conditions — Gastroparesis | interventions — TD-5108

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Velusetrag 5mg (Experimental): Velusetrag 5mg capsules QD (once daily) x 12 weeks
  Interventions: Drug: Velusetrag
- Velusetrag 15mg (Experimental): Velusetrag 15mg capsules QD x 12 weeks
  Interventions: Drug: Velusetrag
- Velusetrag 30mg (Experimental): Velusetrag 30mg capsules QD x 12 weeks
  Interventions: Drug: Velusetrag
- Placebo (Placebo Comparator): Placebo capsules QD x 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Velusetrag
  Other Names: TD-5108
  Arms: Velusetrag 15mg; Velusetrag 30mg; Velusetrag 5mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study 0099 explores the efficacy and safety of multiple doses of velusetrag in the treatment of symptoms in subjects with diabetic or idiopathic gastroparesis. Three dose levels of velusetrag will be evaluated and compared to placebo for approximately 12 weeks of therapy. In addition, the study will be used to evaluate the psychometric properties of the Gastroparesis Rating Scale (GRS), a daily patient-reported outcome (PRO) measure.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of gastroparesis (eg, nausea, early satiety, fullness, bloating, upper abdominal pain, retching or vomiting) for at least 3 months prior to Screening
* Composite score ≥2and <5 on nausea, bloating, feeling excessively full after meals, and not able to finish a normal-sized meal items (on the GCSI-2W) at Screening
* Delayed gastric emptying by either GES (gastric emptying scintigraphy) or GEBT(gastric emptying breath test)
* Upper gastrointestinal obstruction ruled out by endoscopy or other imaging (eg, computed tomography) after the onset of gastroparesis symptoms
* Willing to abstain from prohibited medications, including but not limited to, anticholinergics, acetylcholinesterase antagonists, or promotility medications (eg, metoclopramide, domperidone, prucalopride, erythromycin) for: 24 hours prior to gastric emptying test during Screening, if applicable; 24 hours prior to start of the Baseline period; and during the Baseline Period
* GCSI-24H 7-day mean composite score ≥2.5 and <5 at Day 1

Exclusion Criteria:

* If Type 1 or Type 2 diabetic, a glycosylated hemoglobin (HbA1c) level >11%
* Prior history of gastric surgery, including but not limited to gastrectomy, gastric bypass, gastric banding, pyloroplasty, vagotomy, or fundoplication, which has manipulated the natural anatomy of the stomach
* History of intrapyloric botulinum toxin injection within 3 months of Screening or currently has functioning implantable electric stimulator
* History of alcohol or drug abuse or dependence within the last year prior to Screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
7-day mean GCSI-24H (Gastroparesis Cardinal Symptoms Index) composite score | At Week 4

SECONDARY OUTCOMES:
Gastric emptying half-time | At Week 4
Adverse events | 103 days

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Nguyen, MD, Study Director — Theravance Biopharma

REFERENCES:
- [Derived] Abell TL, Kuo B, Esfandyari T, Pfeifer ND, Grimaldi M, Renzulli C, Tacchi R, Zhou K, Barnes CN, Nguyen DD, Nguyen L, Talley NJ, McCallum R. A randomized, double-blind, placebo-controlled, phase 2b study of the efficacy and safety of velusetrag in subjects with diabetic or idiopathic gastroparesis. Neurogastroenterol Motil. 2023 Apr;35(4):e14523. doi: 10.1111/nmo.14523. Epub 2023 Jan 9. PMID 36624727